CLINICAL TRIAL: NCT00830739
Title: A Multi-Modal Investigation of the Smoking Cessation Medication Varenicline: Dopaminergic Modulation of Reward Processing and Cognitive Control
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909044; 09-DA-N044
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-02-26

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence
Keywords: Smoking Cessation; Dopamine; Cognitive Control; Reward Processing; Varenicline
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Chronic nicotine exposure through cigarette smoking affects the level of the brain chemical dopamine. Smokers who attempt to quit experience lower levels of dopamine, which increases anxiety and triggers nicotine cravings that make quitting more difficult.
* Varenicline (Chantix) is a smoking cessation medication that is designed to reduce nicotine craving and withdrawal by slightly increasing levels of dopamine in the brain. Research has shown that varenicline is a safe, well-tolerated, and effective treatment for nicotine dependence, but researchers are interested in learning more about how it affects the brain and its function. Functional magnetic resonance imaging (fMRI) and electroencephalography (EEG) will help researchers study the brain s response to nicotine and varenicline.

Objectives:

- To explore how varenicline affects brain function and behavioral performance in current smokers and healthy volunteers.

Eligibility:

- Individuals between 18 and 55 years of age who are either current smokers (10 or more cigarettes per day) or healthy nonsmoking volunteers.

Design:

* The study will involve nine testing and research visits over 5 to 6 weeks. The first visit will provide an initial assessment and training on the tasks that will be completed during the study.
* Six testing visits will involve fMRI and EEG measurements of brain activity. Each visit will contain two 2-hour scanning sessions, and each session will involve thinking tests. During these visits, participants will receive varenicline and placebo tablets, and wear nicotine patches and placebo patches that do not contain nicotine. Participants will not be told which tablet or patch they are given. This is a crossover study so all participants eventually get nicotine and placebo, as well as varenicline and placebo.
* Two other visits involve different thinking tasks. These visits will not require fMRI or EEG scans.

DETAILED DESCRIPTION:
Objective. Chronic nicotine exposure is thought to lead to alterations in the dopamine (DA) system that leaves smokers in a hypo-dopaminergic state during periods of abstinence. Varenicline (Chantix), a new efficacious smoking cessation medication, is thought to lead to a modest but sustained increase of DA release thereby reducing nicotine craving and withdrawal. While numerous studies have shown that varenicline is a safe, well-tolerated, and effective pharmacological treatment for nicotine dependence, studies exploring the neurophysiological impact of this drug in the human brain have not been conducted. This protocol will utilize an array of reward processing and cognitive control tasks to explore the effects of subtle DA manipulations (induced by smoking cessation, transdermal nicotine, and varenicline) on brain function and behavioral performance. Brain function will be assessed using functional magnetic resonance imaging (fMRI) and electroencephalography (EEG).

Study Population. There will be two study populations: 1) healthy nicotine-dependent adults who smoke 10 or more cigarettes per day; and 2) healthy non-smoking, non-drug dependent controls. Participants must be generally healthy, right-handed, male or non-pregnant/non-lactating females between the ages of 18-55.

Design. After being medically cleared and giving informed consent, each participant will complete several imaging visits (6 visits, on separate days) before and after taking varenicline. Two of these visits will take place before varenicline administration (baseline), two visits after a two-week varenicline dosing period (post-varenicline), and another two after a two-week placebo-pill period (post-placebo-pill). Each set of two scans will involve the randomized, double blind administration of a nicotine transdermal or placebo patch. fMRI and EEG data will be collected after patch application and will involve several tasks designed to probe brain regions in a corticolimbic circuit that may mediate aspects of reward-processing, learning, attention, goal-directed behaviors, and drug abuse.

Outcome Measures. This study involves assessing neurophysiological and behavior differences between cohorts (smokers vs. non-smokers) and conditions (nicotine vs. placebo-patch; baseline vs. varenicline vs. placebo-pill). The primary outcome measures used to ascertain these differences will be: 1) percentage change in fMRI BOLD signal during performance of cognitive control and reward processing tasks; 2) change in ERP component (e.g., error-related negativity) amplitudes; 3) behavioral measures during task performance including reaction times and error rates; 4) scores on mood, personality, and smoking questionnaires; and 5) variations in genes related to nicotinic receptors and DA functioning.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. between the ages of 18-55.
  2. right-handed.
  3. in good health.
  4. free of active DSM-IV dependence, or dependence in partial remission, on alcohol or any drug except nicotine. Past active dependence is acceptable provided it is at least five years in the past and total time of active dependence did not exceed 4 years. Those with past dependence may not have any current use (past 6 months) of the substance on which they were dependent.
  5. able to abstain from alcohol 24hrs before each of the imaging sessions and able to moderate their caffeine intake 12hrs before each session.

In addition, smokers must:

1. smoke 10 or more cigarettes per day and have smoked for more than 2 years.
2. be able to refrain from smoking for up to 12hrs (at 6 different time points) during the study.
3. be able to tolerate the nicotine patch.

In addition, non-smokers must:

(1) Not have a history of daily cigarette smoking lasting more than a month and no smoking within the past 2 years.

EXCLUSION CRITERIA:

1. are not suitable to undergo an fMRI experiment due to certain implanted devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia.
2. have coagulopathies, history of, current superficial, or deep vein thrombosis, musculoskeletal abnormalities restricting an individual s ability to lie flat for extended periods of time.
3. have HIV or Syphilis.
4. regularly use any prescription, over-the-counter or herbal medication that may alter CNS function, cardiovascular function, or neuronal-vascular coupling.
5. have any current, or a history of, neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, history of significant head trauma, or CNS tumor.
6. have any current, or a history of, major psychiatric disorders, substance-induced psychiatric disorders, suicidal ideations and/or suicide attempts, or currently under antidepressant or antipsychotic medication treatment.
7. are cognitively impaired or learning disabled.
8. have significant cardiovascular or cerebrovascular conditions.
9. have moderate to severe renal impairment.
10. are diabetic.
11. have any other major medical condition that in the view of the investigators would compromise the safety of an individual during participation.
12. pregnant, planning to become pregnant, or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11-25; Study Completion 2013-02-26

PRIMARY OUTCOMES:
To improve understanding of the neural and cognitive consequences of nicotine dependence, nicotine abstinence, and varenicline treatment.

SECONDARY OUTCOMES:
To better understand individual differences that may relate to the effects of nicotine in the brain to improve future smoking cessation treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Aceto MD, Martin BR. Central actions of nicotine. Med Res Rev. 1982 Jan-Mar;2(1):43-62. doi: 10.1002/med.2610020104. No abstract available. PMID 6125634
- [Background] Ahmed SH, Kenny PJ, Koob GF, Markou A. Neurobiological evidence for hedonic allostasis associated with escalating cocaine use. Nat Neurosci. 2002 Jul;5(7):625-6. doi: 10.1038/nn872. PMID 12055635
- [Background] Alain C, McNeely HE, He Y, Christensen BK, West R. Neurophysiological evidence of error-monitoring deficits in patients with schizophrenia. Cereb Cortex. 2002 Aug;12(8):840-6. doi: 10.1093/cercor/12.8.840. PMID 12122032
- [Derived] Lesage E, Aronson SE, Sutherland MT, Ross TJ, Salmeron BJ, Stein EA. Neural Signatures of Cognitive Flexibility and Reward Sensitivity Following Nicotinic Receptor Stimulation in Dependent Smokers: A Randomized Trial. JAMA Psychiatry. 2017 Jun 1;74(6):632-640. doi: 10.1001/jamapsychiatry.2017.0400. PMID 28403383
- [Derived] Sutherland MT, Carroll AJ, Salmeron BJ, Ross TJ, Hong LE, Stein EA. Down-regulation of amygdala and insula functional circuits by varenicline and nicotine in abstinent cigarette smokers. Biol Psychiatry. 2013 Oct 1;74(7):538-46. doi: 10.1016/j.biopsych.2013.01.035. Epub 2013 Mar 15. PMID 23506999